CLINICAL TRIAL: NCT07406035
Title: A Randomized, Placebo- and Active Drug-Controlled, Double-Blind, Multicenter, Parallel-Group Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQH3906 Capsules in the Treatment of Active Psoriatic Arthritis
Brief Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQH3906 Capsules in the Treatment of Active Psoriatic Arthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH3906-II-02
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQH3906 Capsule 24 mg (Experimental): Oral administration daily from Day 1 (D1) to Day 85 (D85) Morning Fasting: 3 Capsules of 8 mg TQH3906
  Interventions: Drug: TQH3906 Capsule
- TQH3906 Capsule 16 mg (Experimental): Oral administration daily from Day 1 (D1) to Day 85 (D85) Morning fasting: 2 capsules of 8 mg TQH3906
  Interventions: Drug: TQH3906 Capsule
- TQH3906 Capsule 0 mg (Placebo Comparator): Oral administration daily from Day 1 (D1) to Day 85 (D85) Morning fasting: 3 placebo capsules of TQH3906
  Interventions: Drug: TQH3906 Placebo Capsule
- Tofacitinib Citrate Tablet 5 mg (Active Comparator): Oral administration daily from Day 1 (D1) to Day 85 (D85):
  Morning fasting: 1 tablet of tofacitinib citrate Administer 1 tablet of Tofacitinib Citrate at bedtime.
  Interventions: Drug: Tofacitinib Citrate Tablet 5 mg

INTERVENTIONS:
Drug: TQH3906 Capsule — TQH3906 is a small-molecule inhibitor of tyrosine kinase.
  Arms: TQH3906 Capsule 16 mg; TQH3906 Capsule 24 mg
Drug: TQH3906 Placebo Capsule — Placebo without drug substance.
  Arms: TQH3906 Capsule 0 mg
Drug: Tofacitinib Citrate Tablet 5 mg — Tofacitinib Citrate Tablets are Janus kinase (JAK) inhibitors.
  Arms: Tofacitinib Citrate Tablet 5 mg

SUMMARY:
This study is a marketing-oriented clinical trial of TQH3906 Capsules. A total of 156 participants are planned to be enrolled, aiming to evaluate the dose-effect relationship of TQH3906 versus placebo in the treatment of active Psoriatic Arthritis (PsA) at Week 12, with the proportion of participants achieving an American College of Rheumatology 20% (ACR20) Improvement Criteria (ACR20) response at Week 12 as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written Informed Consent Form, which must meet the following requirements

  * Be willing to participate in the study and able to sign the informed consent form;
  * Be willing and able to complete all study-specific procedures and visits;
* PsA trial participant disease characteristics

  * Aged 18 to 70 years（inclusive）;
  * BMI ≥ 18 kg/m² at screening; diagnosed with PsA for at least 3 months prior to screening, and meeting the Classification Criteria for Psoriatic Arthritis (CASPAR) at screening;
  * Active arthritis at screening and at baseline (Day 1);
  * Has failed or was intolerant to at least one prior therapy;
  * If receiving a conventional synthetic Disease-Modifying Antirheumatic Drug (csDMARD), trial participants must be on only one DMARD, which must have been administered for at least 3 months prior to screening, with a stable dose for at least 28 days prior to the first dose;
  * If using NSAIDs, the dose must have been stable for at least 14 days before the first dose;
  * If using oral corticosteroids, the dose must have been stable for at least 14 days before the first dose;
  * Topical treatments for plaque psoriasis must have remained stable for at least 14 days before the first dose;
* Women of childbearing potential must agree to use effective contraception during the study and for 6 months after the end of the study; men must agree to use effective contraception during the study and for 6 months after the end of the study

Exclusion Criteria:

* Presence of conditions other than PsA:

  * Presence of non-plaque psoriasis (i.e., guttate, inverse, pustular, erythrodermic, or drug-induced psoriasis) at screening or first dose;
  * Presence of any other autoimmune disease, such as rheumatoid arthritis, systemic lupus erythematosus, etc.;
  * Presence of active (i.e., currently symptomatic) fibromyalgia;
* Other Medical Conditions and Medical History:

  * Trial participants who are pregnant or breastfeeding;
  * Evidence of a serious illness/condition or unstable clinical condition, or localized active infection/infectious disease;
  * Any major surgery performed within 30 days prior to the first dose of study treatment, or any planned surgery during the study;
  * Cancer or a history of cancer or lymphoproliferative disease within the past 5 years;
  * New York Heart Association (NYHA) Class III or IV congestive heart failure, or any recent episode of heart failure resulting in NYHA Class III/IV symptoms; or a history of clinically significant ventricular arrhythmia or arrhythmia requiring continuous antiarrhythmic drug therapy;
  * Uncontrolled hypertension at screening or randomization;
  * History of thrombotic disease within 24 weeks prior to screening; viii. History of acute coronary syndrome and/or any major cerebrovascular disease within 24 weeks prior to screening;
  * Current or recent (within 3 months prior to randomization) gastrointestinal disease that may affect absorption of study treatment, including gastrointestinal surgery;
  * Severe blood loss (> 500 mL) or blood transfusion within 4 weeks prior to randomization;
  * Inability to take oral medication;
  * Inability to undergo venipuncture and/or tolerate venous access;
  * History of substance abuse with inability to abstain or presence of a psychiatric disorder;
  * Any other medical, psychiatric, and/or social reason as determined by medical judgment;
* Prior and concomitant medications: If the trial participant has a history of biologic use, the exclusion criteria specified in the protocol will apply;
* Infection-related:

  * Active tuberculosis identified by chest radiography within 6 months prior to screening; trial participants with a negative chest radiography within 3 months prior to screening are eligible if they meet the protocol requirements;
  * Hepatitis C, hepatitis B, or human immunodeficiency virus (HIV) infection; or syphilis infection requiring treatment;
* Abnormal physical examination or laboratory findings;
* Other:

  * History of any major drug allergy; known allergy to any excipient of the investigational product;
  * Inability to comply with the trial protocol;
  * History of substance abuse with inability to abstain or presence of a psychiatric disorder;
  * Participation in another clinical trial and use of another investigational drug (other than for psoriatic arthritis) within 4 weeks prior to the first dose, based on the date of discontinuation from the previous trial;
  * Planned or previous allogeneic bone marrow transplantation or solid organ transplantation;
  * Any condition that, in the investigator's judgment, poses a serious risk to the safety of the trial participant or affects the participant's ability to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
American College of Rheumatology 20% Improvement Criteria | Day 1, 15, 29, 57, 85
  The proportion of trial participants achieving an ACR20 response at Week 12.

SECONDARY OUTCOMES:
ACR20 in the subgroup of trial participants | Day 1, 15, 29, 57, 85
  The proportion of biologic-naive trial participants in the subgroup who achieved ACR20 response at Week 12.
American College of Rheumatology 50 (ACR50) | Day 1, 15, 29, 57, 85
  ACR50 response rate
American College of Rheumatology 70 (ACR70) | Day 1, 15, 29, 57, 85
  ACR70 response rate
Psoriasis Area and Severity Index (PASI) 75 | Day 1, 15, 29, 57, 85
  PASI 75 response rate
Psoriasis Area and Severity Index 90 | Day 1, 15, 29, 57, 85
  PASI 90 response rate
Numbers of subjects with incidence of adverse Event (AE), serious Adverse Event (SAE), adverse event leading to study discontinuation, adverse event of special interest (AESI) | From the time trial participants sign the informed consent form to 28 days after the last dose
  Numbers of subjects with incidence rates of Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events Leading to Study Discontinuation, and Adverse Events of Special Interest (AESIs)
Time to Peak Concentration (Tmax) | Up to day 85
  Evaluation of the Time to Peak Concentration (Tmax) of TQH3906 in participants with Psoriatic Arthritis after oral administration.
Peak Concentration (Cmax) | Up to day 85
  Evaluation of the Peak Concentration (Cmax) of TQH3906 in Participants with Psoriatic Arthritis After Oral Administration
Plasma Clearance (CL/F) | Up to day 85
  Evaluation of the Plasma Clearance (CL/F) of TQH3906 in Participants with Psoriatic Arthritis After Oral Administration.
Plasma Elimination Half-Life (t₁/₂) | Up to day 85
  Evaluation of the Plasma Elimination Half-Life (t₁/₂) of TQH3906 in Participants with Psoriatic Arthritis After Oral Administration.
Trough Concentration at Steady State (Cmin, ss) | Up to day 85
  Evaluation of the Trough Concentration at Steady State (Cmin, ss) of TQH3906 in Participants with Psoriatic Arthritis After Oral Administration.
Degree of Fluctuation (DF) | Up to day 85
  Evaluation of the Degree of Fluctuation (DF) of TQH3906 in Participants with Psoriatic Arthritis After Oral Administration.
Evaluation of Interleukin (IL) Levels in Participants with Psoriatic Arthritis Treated with TQH3906 | Blood samples were collected within 1 hour before dosing at Baseline, Weeks 2, 4, 8, and 12
  Evaluation of Interleukin (IL) Levels in Participants with Psoriatic Arthritis Treated with TQH3906
Evaluation of Defensin Levels in Participants with Psoriatic Arthritis Treated with TQH3906 | Blood samples were collected within 1 hour before dosing at Baseline, Weeks 2, 4, 8, and 12
  Evaluation of Defensin Levels in Participants with Psoriatic Arthritis Treated with TQH3906

CONTACTS AND LOCATIONS:
Locations (42):
- China (42):
  - Bozhou People's Hospital, Bozhou, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, Third Military Medical University (Army Medical University), Chongqing, Chongqing Municipality
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Bao Ding NO.1 Central, Baoding, Hebei
  - Hebei Cangzhou Hospital of Integrated Traditional Chinese Medicine and Western Medicine, Cangzhou, Hebei
  - Kaifeng People's Hospital, Kaifeng, Henan
  - Luoyang Orthopedic-Traumatological Hospital Of Henan Province(Henan Provincial Orthopedic Hospital), Luoyang, Henan
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of CM, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Central Hospital of Shaoyang, Shaoyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Jiangsu Peopince Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Yancheng No.1 People's Hospital, Yancheng, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The second hospital of dalian medical university, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Weifang People'S Hospital, Weifang, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Deyang People's Hospital, Deyang, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Li HuiLi Hospital, Ningbo, Zhejiang